CLINICAL TRIAL: NCT05084664
Title: Effect of Premodulated Current Versus Diadynamic Current On the Management of Tennis Elbow.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Emad Eldin Mohamed, lecturer (header of basic science department), October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 897
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): premodulated current
  Interventions: Device: electrical stimulation
- group B (Experimental): diadynamic current
  Interventions: Device: electrical stimulation

INTERVENTIONS:
Device: electrical stimulation — premodulated current+ exercises
  Arms: group A
Device: electrical stimulation — diadynamic current+ exercises
  Arms: group B

SUMMARY:
104 patients with unilateral tennis elbow from both genders (57 females and 43 males) referred by orthopaedist with age ranged between 20 and 60 years.

DETAILED DESCRIPTION:
hey were recruited in the study from October 2020 to September 2021 and allocated randomly into two groups. Group A received premodulated current in addition to exercises, and group B received diadynamic current with the same exercises. Each patient signed the informed consent form approved by the faculty of physical therapy, October 6 university, Egypt and prospectively registered (Clinical Trials.gov, Identifier NCT03338283). Patients was selected according to the following criteria.

Inclusive criteria

* Patients suffer from pain at the lateral part of the elbow and radiated to the forearm with tenderness increasing on pressure on the lateral epicondyle and on resistance of hand extension
* lasting of the symptoms for 3 months
* no previous physiotherapy interventions.

Exclusive criteria

Internal or external fixation

* arthritis of elbow
* contraindications to electrotherapy like pacemaker, dermatological skin disease, epilepsy, abnormal sensation, and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from pain at the lateral part of the elbow and radiated to the forearm with tenderness increasing on pressure on the lateral epicondyle and on resistance of hand extension
* lasting of the symptoms for 3 months
* previous physiotherapy interventions.

Exclusion Criteria:

* Internal or external fixation
* arthritis of elbow
* contraindications to electrotherapy like pacemaker, dermatological skin disease, epilepsy, abnormal sensation, and pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
baseline hydraulic hand dynamometer | 6 weeks
  grip strength measurement (200 lb.90 kg Capacity)
Patient-Rated Tennis Elbow Evaluation (PRTEE) | 6 weeks
  pain and functional measurement (The maximum score is 50 for the pain subscale and 100 for the function subscale)
baseline hydraulic pinch gauge | 6 weeks
  pinch measurement (50 lb.22.5 kg Capacity)

CONTACTS AND LOCATIONS:
Locations (1):
- Bassam, Qaliubia, Egypt

IPD SHARING:
Plan to Share IPD: No